CLINICAL TRIAL: NCT02330783
Title: A Randomized, Open-label, Multi-center Phase II Study to Compare Bevacizumab Plus Sorafenib Versus Sorafenib for the Third-line Treatment of Patients With Metastatic Renal Cell Carcinoma
Brief Title: Efficacy and Safety of Bevacizumab Plus Sorafenib for the Third-line Treatment in Metastatic Renal Cancer Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Jun Guo, Director of department of renal cancer and melanoma, Peking University Cancer Hospital & Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BCH-RCC-141201
Record Dates: First submitted 2014-12-29; First posted 2015-01-05 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Metastatic Renal Cell Carcinoma
Keywords: Metastatic Renal Cell Carcinoma; Third-line treatment; Sorafenib; Bevacizumab
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Bevacizumab; Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bevacizumab plus Sorafenib (Experimental): Bevacizumab 5mg/kg Q2w Sorafenib 400mg Bid
  Interventions: Drug: Bevacizumab; Drug: Sorafenib
- Sorafenib (Active Comparator): Sorafenib 400mg Bid
  Interventions: Drug: Sorafenib

INTERVENTIONS:
Drug: Bevacizumab — 5mg/kg by intravenous (IV) infusion every two weeks of each 4-week cycle (dose was based on patient's weight at screening and remained the same throughout study)
  Other Names: Avstin
  Arms: Bevacizumab plus Sorafenib
Drug: Sorafenib — 400mg twice daily by oral of each 4-week cycle
  Other Names: Nexavar

SUMMARY:
There is no standard treatment in patients with renal cell carcinoma that was previously treated with VEGF targeted therapies and mTOR inhibitors.So investigators conducted a randomized, open-label, multi-center phase II study to compare bevacizumab plus sorafenib versus sorafenib for the third-line treatment of patients with Metastatic renal cell carcinoma.

DETAILED DESCRIPTION:
Therapies targeting VEGF and mTOR signalling pathways represent standard first-line and second-line treatment options for patients with metastatic renal cell carcinoma. There is no standard treatment in patients with renal cell carcinoma that was previously treated with VEGF targeted therapies and mTOR inhibitors.To the best of the investigators knowledge, GOLD study is the first phase 3 trial in the third-line setting after both VEGF-inhibitor and mTOR-inhibitor drugs.From this study,Sorafenib may be option for the third-line treatment.The Best trial demonstrated that Bevacizumab/sorafenib had best efficacy in advance renal cancer canrcinoma and the VEGF/VEGFR co-inhibition strategy may warrant further investigation possibly with more selective VEGFR inhibitors.So investigators conducted a randomized, open-label, multi-center phase II study to compare bevacizumab plus sorafenib versus sorafenib for the third-line treatment of patients with Metastatic renal cell carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Age≥18 years, ≤75 years, male or female
* Advanced renal cellcarcinoma is diagnosed histologically or pathologically

  * 1st line treatment of Sunitinib and 2nd line treatment of Everolimus and no more systemic anti-angiogenesis targeted drug therapy
  * Have at least one measurable tumor lesion (Response Evaluation Criteria In Solid Tumors)
  * Eastern Cooperative Oncology Group（ECOG) performance scale is 0 or 1
  * The expected life span is ≥12 weeks
  * No contraindications for chemotherapy, with enough liver function and renal function and normal ECG recording Peripheral hemogram: neutrophil≥1.5×109/L, Plt≥100×109/L, Hgb≥90g/L Renal function: serum creatinine≤1.5 folds the upper limit of normal (ULN) For patients with non-metastatic liver dysfunction:alanine aminotransferase and aspartate aminotransferase≤2.5 ULN, For patients with metastatic liver dysfunction: alanine aminotransferase and aspartate aminotransferase≤5 ULN
  * The patients participate voluntarily and have signed the informed consent form

Exclusion Criteria:

* Pregnant and lactating women, or female patients of child-bearing age without taking contraceptive measures

  * Patients with severe acute infection without being controlled effectively or having pyogenic and chronic infections with persistently unhealed wounds
  * Past history of serious heart diseases, including: cardiac function classification ≥NYHA class II, unstable angina pectoris, myocardial infarction, arrhythmia requiring anti-arrhythmic drug therapy (excluding β-blockers or digoxin), and uncontrolled hypertension
  * Patients with a history of HIV infection or active phase of chronic hepatitis B/C
  * negative imaging examination result 4 weeks prior to enrollment)
  * Epilepsy patients requiring drug therapy (e.g. steroids or antiepileptic drugs)
  * A history of allogeneic organ transplantation
  * Patients with evidence of hemorrhagic constitution or a past history of hemorrhage
  * Patients currently receiving renal dialysis
  * Past or present concomitant tumors with the primary lesions or histological characteristics different from the tumors evaluated in this study, excluding other tumor cured longer than 3 years before enrollment
  * Patients participating in other clinical trials simultaneously
  * Other conditions unsatisfying the inclusion criteria in the investigator's opinions

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2014-12; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
progress-free survival,PFS | 2 years
  Time from enrollment to the dates of disease progression,death from any cause or last tumor assessment reported between date of first patient enrollment until 31 December 2017 cut of date

SECONDARY OUTCOMES:
overall survival,OS | 3 years
  Time from enrollment to the dates of death from any cause or last follow up reported between date of first patient enrollment until 31 December 2017 cut of date
Safety: adverse events | 1 years
  adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Jun Guo, MD,PHD, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (4):
- China (4):
  - Sun Yat-sen university cancer center, Guangzhou, Guangdong
  - Peking University First Hospital, Beijing
  - Beijing Cancer Hospital, Beijing
  - Cancer Hospital, Fudan University, Shanghai

REFERENCES:
- [Background] Motzer RJ, Porta C, Vogelzang NJ, Sternberg CN, Szczylik C, Zolnierek J, Kollmannsberger C, Rha SY, Bjarnason GA, Melichar B, De Giorgi U, Grunwald V, Davis ID, Lee JL, Esteban E, Urbanowitz G, Cai C, Squires M, Marker M, Shi MM, Escudier B. Dovitinib versus sorafenib for third-line targeted treatment of patients with metastatic renal cell carcinoma: an open-label, randomised phase 3 trial. Lancet Oncol. 2014 Mar;15(3):286-96. doi: 10.1016/S1470-2045(14)70030-0. Epub 2014 Feb 17. PMID 24556040
- [Background] Sosman JA, Puzanov I, Atkins MB. Opportunities and obstacles to combination targeted therapy in renal cell cancer. Clin Cancer Res. 2007 Jan 15;13(2 Pt 2):764s-769s. doi: 10.1158/1078-0432.CCR-06-1975. PMID 17255307
- [Background] Azad NS, Posadas EM, Kwitkowski VE, Steinberg SM, Jain L, Annunziata CM, Minasian L, Sarosy G, Kotz HL, Premkumar A, Cao L, McNally D, Chow C, Chen HX, Wright JJ, Figg WD, Kohn EC. Combination targeted therapy with sorafenib and bevacizumab results in enhanced toxicity and antitumor activity. J Clin Oncol. 2008 Aug 1;26(22):3709-14. doi: 10.1200/JCO.2007.10.8332. PMID 18669456
- [Background] Pal SK, Vogelzang NJ. Sequential treatment strategies and combination therapy regimens in metastatic renal cell carcinoma. Clin Adv Hematol Oncol. 2013 Mar;11(3):146-55. PMID 23598982